CLINICAL TRIAL: NCT00844831
Title: Effects of Lubiprostone on Small Bowel and Colonic Bacteria: A Correlation Study With Segmental and Whole Gut Transit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 285.09
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Constipation
Keywords: Constipation; small intestinal bacterial overgrowth; stool bacteria
MeSH Terms: conditions — Constipation | interventions — Lubiprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with lubiprostone (Experimental): Subjects receive lubiprostone and bacteria is measured before and after
  Interventions: Drug: Lubiprostone

INTERVENTIONS:
Drug: Lubiprostone — 24 mcg bid for 28 days
  Other Names: Amitiza

SUMMARY:
Patients with constipation often have bloating and abdominal distension. It is unclear if this is related to intestinal bacteria. Hypothesis: treatment for constipation may reduce small bowel and colon bacteria colonization, a change in the balance of stool microorganisms, and improve the symptoms of dyspepsia and constipation.

DETAILED DESCRIPTION:
This is an open-label study to collect data on upper and lower GI symptoms, hydrogen breath test, stool PCR, and serum before and after 4 weeks of lubiprostone 24 mcg by mouth twice a day for 4 weeks.

ELIGIBILITY:
Inclusion Criteria: Functional constipation by Rome III criteria

Exclusion Criteria:

1. History of esophageal or gastric surgery (including vagotomy, antireflux, and obesity surgery)
2. History of small bowel or colon resection (excluding appendectomy and cholecystectomy)
3. History of gastric outlet, small bowel, or colon obstruction
4. History of surgery for small bowel adhesion lysis
5. History of surgery for gastroparesis
6. Diagnosis of diabetes requiring daily medications
7. Diagnosis of connective tissue d/o (including scleroderma, lupus, mixed connective tissue disorder)
8. Diagnosis of neuromuscular disorder (including multiple sclerosis, Parkinson, muscular dystrophy, dysautonomia, dystonia)
9. Disorders of small bowel pseudo-obstruction or dumping syndrome
10. Untreated or poorly controlled hypothyroidism
11. Taking an opiate medication daily
12. Taking a medication daily that can cause constipation (calcium channel blocker, anticholinergic, iron supplements, etc.)
13. Active cancer being treated
14. History of significant liver, kidney, cardiac disease that may interfere with study compliance
15. Known allergy or side effects to lubiprostone
16. Non-ambulatory patients: bed-ridden, nursing home resident, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Wo, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from outpatient clinics and advertisement
Pre-assignment Details: Study consisted of a 4-week run-in period to wash out prior therapy for constipation. Subjects may withdraw if they can not stay off their medications for constipation.
Period: Overall Study
Arm/Group | Lubiprostone Open Label
Started | 25
Completed | 19
Not Completed | 6
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lubiprostone Open Label
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Presence of Small Intestinal Bacterial Overgrowth
Description: Percent of patients with bacterial overgrowth before and after treatment.
Time Frame: 28 days
Population: ITT
Measure: Count of Participants; unit: Participants
Groups:
- Before Open Label Lubiprostone: Before 4-wk treatment period with open label lubiprostone 24 mcg tablet po twice daily.
- After Open Label Treatment: After 4-wk treatment period with open label lubiprostone 24 mcg tablet po twice daily
Arm/Group | Before Open Label Lubiprostone | After Open Label Treatment
Number analyzed (Participants) | 19 | 19
Participants | 8 | 9
Statistical Analysis 1: Comparison: Before Open Label Lubiprostone vs After Open Label Treatment; Test type: Superiority; p = 0.75, t-test, 2 sided

2. Secondary Outcome: Small Bowel and Colon Transit Time by SmartPill® Transit Study
Time Frame: 28 days
Population: We were unable to obtain the smart pills for this section of the protocol.
Arm/Group | Treatment With Lubiprostone
Number analyzed (Participants) | 0

3. Secondary Outcome: Small Intestinal Bacterial Overgrowth (SIBO)
Description: SIBO was measured before and after treatment.
Time Frame: 28 days
Measure: Number; unit: participants
Groups:
- Before Open Label Lubiprostone: Bacteria is measured before Lubiprostone: 24 mcg bid for 28 days
- After Open Label Treatment: Subjects receive lubiprostone and bacteria is measured after Lubiprostone: 24 mcg bid for 28 days
Arm/Group | Before Open Label Lubiprostone | After Open Label Treatment
Number analyzed (Participants) | 19 | 19
participants | 8 | 9
Statistical Analysis 1: Comparison: Before Open Label Lubiprostone vs After Open Label Treatment; Test type: Other; p = .9, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Groups:
- Lubiprostone Open Label: 4-wk treatment period with open label lubiprostone 24 mcg tablet po twice daily
Arm/Group | Lubiprostone Open Label
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lubiprostone Open Label (N=25)
Transient ischemic attack (Nervous system disorders) | 1 (1) — One male subject was withdrawn due to developing a transient ischemia attack during the treatment period, and subsequent testing revealed carotid artery atherosclerotic disease. This event was considered unrelated to the study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No